CLINICAL TRIAL: NCT03170479
Title: Developmental Screening and Nutritional Intervention of Severe Acute Malnourished Children in Southern Punjab, Pakistan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of the Punjab (Other)
Responsible Party: Principal Investigator, Dr. Javeria Saleem, Principal Investigator, University of the Punjab
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UPunjab
Record Dates: First submitted 2016-10-16; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Malnutrition in Children
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RUTF with Vitamin D (Experimental): Two groups (arms) of malnourished children will be made, one study and one control group; Experimental arm will use RUTF and two mega doses of 200,000 IU vitamin D randomly first after 15 days of enrollment and second after 15 days of first dose.
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Ready to Use Therapeutic Food (RUTF)
- RUTF with Placebo (Placebo Comparator): Placebo arm will receive Ready to Use Therapeutic Food (RUTF) and extra virgin olive oil as Placebo.
  Interventions: Dietary Supplement: Ready to Use Therapeutic Food (RUTF)

INTERVENTIONS:
Dietary Supplement: Vitamin D — Two doses of Vitamin D supplementation in ampoules form (ED3) were procured. Ampoule contains Cholecalciferol in 200,000 IU both for oral and intra muscular use.
  Arms: RUTF with Vitamin D
Dietary Supplement: Ready to Use Therapeutic Food (RUTF) — RUTF is recommended by WHO for sever malnourished children in community settings as a therapeutic diet. The quantity depends upon the child body weight.

SUMMARY:
i. To examine the impact of malnutrition on development quotient of children

ii. To determine the effectiveness of Ready to Use Therapeutic Food (RUTF) in improving the development quotient of severe acute malnourished children under five year of age.

iii. To investigate the outcome of Vitamin D therapeutic doses intervention with RUTF rehabilitation on growth and development of malnourished children.

DETAILED DESCRIPTION:
1. Research Instrument: For Development quotient Denver 2 screening form and tools will be used. Follow up of patients for three months and for recording of their weight Community management of acute malnutrition forms will be used. Denver screening tool will be used for child development quotient covering all areas of development, fine motor, gross motor, language and personal social contact.
2. Research Settings: The study will be conducted in Dera Ghazi Khan division at, Basic Health Units (BHU).
3. Study design: Randomized Controlled Trial.
4. Data Collection: Lady Health Visitors (LHWs) will screen the children aged 6 months to 59 months in their community and will refer the severely malnourished children to Outpatient Therapeutic Programs (OTPs).Two groups of malnourished children will be made one study and one control group; one group will be treated with RUTF and extra virgin olive oil as placebo. Other will with RUTF and two mega doses of Vitamin D randomly, first after 15 days of enrollment and second after 15 days of first dose.

ELIGIBILITY:
Inclusion Criteria

* All the selected children of Severe uncomplicated acute malnutrition of concerned age group whose parents or guardians have give written consent for the study
* Mid Upper Arm Circumference (MUAC) less than 11.5 cm or Weight For Height (WFH) less then minus 3 standard deviation.

Exclusion Criteria

* Children above the concerned age group
* Refusal of parents for taking part in the study.
* Child having Severe Acute Malnutrition (SAM) with complications have loss of appetite, lower respiratory tract infection indicated by chest in drawing, severe vomiting.
* Temperature greater then 39°C or hypothermia less then 35°C, very pale, oedema, unconsciousness.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 185 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Weight gain in children | 2 Months
  More than 15% weight gain from enrollment date

SECONDARY OUTCOMES:
Developmental Milestones of children | 2 Months
  Normal or delayed development using Denver Developmental Screening Tool 2 (DDST2)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Z Zakar, PhD, Study Director — University of the Punjab

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Saleem J, Zakar R, Zakar MZ, Belay M, Rowe M, Timms PM, Scragg R, Martineau AR. High-dose vitamin D3 in the treatment of severe acute malnutrition: a multicenter double-blind randomized controlled trial. Am J Clin Nutr. 2018 May 1;107(5):725-733. doi: 10.1093/ajcn/nqy027. PMID 29722846